CLINICAL TRIAL: NCT00743626
Title: Evaluation of the Role of Human Papillomavirus Testing and p16 Expression in the Management of Patients Undergoing Cervical Cancer Screening
Brief Title: Pap Smear Research Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pap Smear Study
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Cervical Cancer
Keywords: Pap test; HPV; Healthy patients screened for cervical cancer tests.
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Papanicolaou Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Healthy patients screened for cervical cancer
  Interventions: Other: Diagnostic cervical cancer screening tests (Pap smear, HPV and/or p16)

INTERVENTIONS:
Other: Diagnostic cervical cancer screening tests (Pap smear, HPV and/or p16) — If positive (Pap smear, HPV and/or p16) patients will be scheduled for 3 colposcopy follow up visits (1,12,18 months)

SUMMARY:
The principal hypothesis of this study is that HPV testing and/or p16 testing, either alone or in combination or associated with a Pap smear, will demonstrate greater specificity for clinically significant precancerous disease than will a Pap smear alone and that these tests will be of comparable or superior sensitivity than the Pap smear.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Ability to speak and clearly understand English
* Female patients

Exclusion Criteria:

* No previous history of Cervical Cancer Treatment(LEEP,Laser,Cone etc.)
* Women who have had Pap smears within the previous 10 months
* Women under the age of 18.
* Women who are pregnant.
* Inability to give informed consent in English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1712 (Actual)
Dates: Start 2006-12 (Actual); Primary Completion 2008-08 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To provide cervical cancer screening (Pap smear, HPV test and/or p16 tests) to determine whether further intervention (colposcopy) is required | 1st visit, 12 months, 18 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Joan K Murphy, MD,FRCSC, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network - Toronto Western Hospital, Toronto, Ontario, Canada